CLINICAL TRIAL: NCT06104436
Title: The Effects of an Individualized Music Playlist Based on the ISOPrinciple for the Immediate De-escalation of Agitation in People With Dementia: a Randomized Controlled Trial
Brief Title: Individualized Music Playlist Based on ISO Principle for De-escalation of Agitation in Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A0047147
Record Dates: First submitted 2023-09-28; First posted 2023-10-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Dementia
Keywords: Dementia; Agitation; Music
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized music playlist (Experimental): Composed of preferred music genres sequenced according to the ISO-Principle in addition to usual care.
  Interventions: Behavioral: Individualized music playlist; Behavioral: Usual care
- Preferred music (Active Comparator): Preferred music genres played in random sequence in addition to usual care.
  Interventions: Behavioral: Preferred music; Behavioral: Usual care
- Treatment as usual (Sham Comparator): Usual care for agitation management.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Individualized music playlist — Individualized music playlist composed of preferred music genres sequenced according to the ISO-Principle. It will be played at the state of agitation.
  Arms: Individualized music playlist
Behavioral: Preferred music — Preferred music is composed of the genres selected by the participants, and to be played at random sequence.
  Arms: Preferred music
Behavioral: Usual care — Usual technique for calming agitated older adults with dementia

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of an Individualized Music Playlist (InMP) composed of preferred music genres sequenced according to the ISO-Principle, for the immediate de-escalation of agitation in dementia, compared with preferred music (PM) and treatment as usual (TAU).

DETAILED DESCRIPTION:
1. Study design

   - Randomized controlled trial
2. Participants

   - Eighty-one older adults living with dementia and demonstrate significant agitation
3. Setting:

   - Residential care home
4. Intervention

   - Individualized music listening intervention played with an iPad and a wireless neckband speaker for 30 minutes when agitation begins in addition to usual care.
5. Comparison conditions

   * Preferred music listening group: Preferred music listening played with an iPad and a wireless neckband speaker for 30 minutes when agitation begins in addition to usual care.
   * Usual care group: usual care
6. Outcomes

   * Level of agitation measured with the Pittsburgh Agitation Scale
   * Intensity of agitation measured with the Positive and Negative Syndrome Scale - Excited Component
   * Agitation occurrence frequency measured with Cohen-Mansfield Agitation Inventory
   * Distress of formal caregivers related to agitation measured with Neuropsychiatric Inventory
7. Focus group interviews with the care staff will be conducted as a process evaluation for identifying the potential facilitators and barriers related to implementation.

ELIGIBILITY:
Inclusion Criteria:

* residents in long-term care facilities
* diagnosed with any type of dementia
* presented with significant agitation

Exclusion Criteria:

* had been admitted to the facility for less than three months
* are participating in other studies or experimental therapies
* have a comorbid psychiatric illness
* have physical illness that prevents them from listening to music

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of agitation | 6 weeks
  Positive and Negative Syndrome Scale - Excitatory Component will be used for assessing the level of agitation. It consists of 5 items: excitement, tension, hostility, uncooperativeness, and poor impulse control. The 5 items from the PANSS-EC are rated from 1 (not present) to 7 (extremely severe); scores range from 5 to 35; mean scores ≥ 20 clinically correspond to severe agitation.
Intensity of agitation | 6 weeks
  Pittsburgh Agitation Scale will be used to assess the intensity of agitation. It is a brief measure of agitation that measures the severity of agitation in four general categories: aberrant vocalisation, motor agitation, aggressiveness and resisting care, on a scale from 0 (not present) to 4 (highest level).
Agitation status | 6 weeks
  Behavioural Activity Rating Scale will be used to assess the agitation status. It contains a single-item question consisting of seven categories: 1=difficult or unable to rouse; 2=asleep, but responds normally to verbal or physical contact; 3=drowsy, appears sedated; 4=quiet and awake (normal level of activity); 5=signs of overt (physical or verbal) activity, calms down with instruction; 6=extremely or continuously active, not requiring restraint; 7=violent, requires restraint.

SECONDARY OUTCOMES:
Agitation occurrence | 6 weeks
  Cohen-Mansfield Agitation Inventory will be used to assess the agitation occurence. A total CMAI score is obtained by summing all the individual items, giving a range from 29 to 203. A total score of >45 is usually regarded as clinically significant agitation.
Emotional or psychological distress of carer | 6 weeks
  Neuropsychiatry Inventory Questionnaire will be used to assess the distress of caregivers. Caregiver distress is rated for each positive neuropsychiatric symptom domain on a scale anchored by scores from 0 to 5 points (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=very severe distress), giving a maximum score of 60.

OTHER OUTCOMES:
Challenges and enablers in the implementation of the intervention | 6 weeks
  Semi-structured focus group interviews with the carers will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Sze Ki Cheung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No